CLINICAL TRIAL: NCT05728307
Title: Evaluating the Clinical Impact and Cost-effectiveness of a Wireless Vital Sign Monitor for Hospitalized Newborns in Kenya
Brief Title: Post-market Observation of a Wireless Vital Sign Monitor for Hospitalized Newborns in Kenya
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assumpta Solome Nantume (Industry)
Collaborators: Academic Model Providing Access to Healthcare (AMPATH) (Other); DLR German Aerospace Center (Other)
Responsible Party: Sponsor-Investigator, Assumpta Solome Nantume, Research & Evaluation Lead, Neopenda, PBC
Organization: Neopenda, PBC (Industry)
Other Study IDs: FAN:0003994
Record Dates: First submitted 2023-01-24; First posted 2023-02-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Newborn Complication; Newborn Morbidity
Keywords: Vital signs monitoring; Health technology; Medical device; Wearable device

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention Group: The intervention group consists of patients admitted to the 4 neonatal subunits where neoGuard was installed: the preterm units (category A and category B), and the high dependence units (HDU-1 and HDU-2).
  Interventions: Device: neoGuard vital signs monitor
- Comparison Group: The comparison group consists patients admitted 4 subunits where neoGuard was not installed: the neonatal intensive care unit (NICU), the KMC/category C room, the isolation room and the stable full-term room. These subunits will receive the standard-of-care/current practice, which consists of either a bedside cardiac monitor or intermittent monitoring every 3 hours using manual equipment such as hand-held pulse oximeters for pulse rate and oxygen saturation, digital axillary thermometers for temperature, and manual counting of breaths for respiratory rate.

INTERVENTIONS:
Device: neoGuard vital signs monitor — The neoGuard device is a 4-in-1 wearable vital signs monitor developed by Neopenda, PBC (Chicago, Illinois). The system is designed to continuously measure temperature, pulse rate (PR), respiratory rate (RR) and blood oxygen saturation (SpO2). It contains two non-invasive sensors: an optical reflectance pulse oximeter and a digital temperature sensor. These sensors measure signals from the surface of the patient's skin, and algorithms within the device calculate the pulse rate, respiratory rate, SpO2 and temperature.
  The device is made of medical grade polyetherimide plastic and can be worn on the forehead through an adjustable band. The PR, RR, temperature and SpO2 data are collected, recorded and transmitted via Bluetooth Low Energy (BLE) to a tablet which can be placed within a range of 20-30 meter distance. The neoGuard technology has received CE mark certification and is also registered with the Kenya Pharmacy and Poisons Board (KPPB).
  Groups: Intervention Group

SUMMARY:
The goal of this study is to measure the clinical impact and cost-effectiveness of a wireless vital signs monitor, neoGuard, for hospitalized newborns at a tertiary healthcare facility in Kenya. The main questions it aims to answer are:

1. Does the neoGuard vital signs monitor detect meaningful vital sign changes in hospitalized newborns?
2. Does the neoGuard vital signs monitor generate valid signals to trigger a timely response from nurses?
3. Is the neoGuard vital signs monitor associated with improved patient outcomes and lower mortality?
4. What is the cost-effectiveness of the neoGuard vital signs monitor in comparison to the standard-of-care monitoring system? Participants will be enrolled within the first 24 hours of admission and monitored for a period of 7 consecutive days or until they are discharged (whichever comes sooner).

The study will consist of an intervention group and a comparison group. Researchers will compare nurses' response time to patients in distress, newborn complication rates and treatment outcomes between the two groups.

DETAILED DESCRIPTION:
This is an interrupted time series study conducted at the Moi Teaching and Referral Hospital (MTRH) neonatal ward between April 2022 and June 2023. Our study participants comprise of newborn patients admitted at MTRH during that period. The MTRH neonatal ward is arranged in 8 sub-units which comprise our comparison sub-groups. Newborns admitted from April-November 2022 comprise the pre-intervention arm and are not exposed to neoGuard, but receive existing standard-of-care vital sign monitoring.

In December 2022, neoGuard was installed in 4 sub-units (intervention group), while the remaining 4 sub-units (comparison group) continued to use standard-of-care monitoring.

The measurement of effectiveness will be performed at three levels: (1) device's ability to detect abnormal physiological signals and provide alerts/alarms that notify the nurses to check on a patient's status and; (2) alarms/alerts from level one that resulted in a necessary intervention being administered to the patient (valid alarms), versus all the alarms/alerts that did not necessitate an intervention (invalid alarms); (3) the month-to-month difference in newborn complication rates and treatment outcomes between the intervention group and comparison group.

Medical staff who interact with neoGuard will participate in user surveys at the end of the intervention period to capture user experience and perceptions on feasibility and sustainability.

ELIGIBILITY:
Inclusion Criteria:

* Must be admitted to one of the subunits assigned to receive the intervention (i.e., APU category A or B, the HDU-1 or HDU-2)
* The newborn's parent/guardian must provide informed consent to use the neoGuard system on their newborn.

Exclusion Criteria:

* Assessed to have congenital anomalies that are incompatible with life
* Receiving palliative care
* Patients undergoing phototherapy
* Those with open head injuries/lacerations
* Those receiving treatment that might interfere with application of the neoGuard device

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population consists of newborns aged 0-28 days admitted to the neonatal ward at MTRH between April 2022-June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Nurse's response time to patients in distress | Captured in real time through monitor logs, within a few seconds to minutes of the event
  The time elapsed (in seconds) between the neoGuard alarm being triggered (distress signal) and the nurse attending to the patient
Percentage of actionable alarms | Measured over a maximum period of 7 days for each patient
  The overall proportion of alarms that are indicative of a true physiological change (distress signal) resulting in an intervention or treatment of the patient

SECONDARY OUTCOMES:
Incidence of patient complications | Through study completion, across 64 weeks
  Bi-weekly change in the incidence of patient complications
In-hospital mortality | Through study completion, across 16 months
  Month-to-month change in the incidence of in-hospital mortality
Frequency of key interventions | Through study completion, across 16 months
  Month-to-month change in the frequency of key interventions administered (i.e., cPAP, supplemental oxygen, mechanical ventilation, antibiotic therapy)

OTHER OUTCOMES:
Qualitative feedback from health providers | Once, at study completion
  Nurses will be surveyed about their experience and perceptions of the technology

CONTACTS AND LOCATIONS:
Overall Officials: Festus Njuguna, MMed, Principal Investigator — Moi Teaching and Referral Hospital/Moi University
Locations (1):
- Moi Teaching and Referral Hospital, Eldoret, Kenya

IPD SHARING:
Plan to Share IPD: No